CLINICAL TRIAL: NCT06617117
Title: Dynamic Acute Responses of Different Intensity-dependent Exercises on the Autonomic and Vascular Systems in People with Coronary Artery Disease
Brief Title: Central Vs Brachial BP, Exercise, and Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BRAVE HEARTS
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: Central blood pressure; Brachial blood pressure; acute exercise; exercise intensity; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Parallel group crossover randomized trial
Masking Description: Outcomes will be assessed by the same experts in every time point. Participants and evaluators will be blinded until arrival of the participant for the first experimental condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate-intensity combined exercise (Experimental): A one-hour exercise session of moderate-intensity structured as follows: a warm-up (10 min), aerobic exercise (20 min), followed by a circuit resistance exercise (20 min), concluded with passive stretching cool down (10 min).
  Interventions: Other: Moderate-intensity combined exercise
- High-intensity combined exercise (Experimental): A one-hour exercise session of high-intensity structured as follows: a warm-up (10 min), aerobic exercise (20 min), followed by a circuit resistance exercise (20 min), concluded with passive stretching cool down (10 min).
  Interventions: Other: High-intensity combined exercise

INTERVENTIONS:
Other: High-intensity combined exercise — The main part consisted of interval cycling exercise, comprising 5x2 min at the second ventilatory threshold interspersed with 4x2 min at the first ventilatory threshold, followed by 2-min unloading pedalling. Subsequently, participants completed resistance exercises (2 sets of 12 repetitions), targeting the same muscle groups of the moderate-intensity exercise, at an intensity of 80% of their 1 repetition maximum.
  Arms: High-intensity combined exercise
Other: Moderate-intensity combined exercise — The main part of the exercise session consisted of an 18-min cycling continuous aerobic exercise at the first ventilatory threshold, followed by 2-min of unloading cycling. Subsequently, participants engaged in resistance exercises - 2 sets of 12 repetitions at 60% of their one repetition maximum. These resistance exercises were part of a machine-assisted circuit training program, encompassing Chest Press, Leg Curl, Low Row, Leg Press, Lat Pull-down, and Leg Extension.
  Arms: Moderate-intensity combined exercise

SUMMARY:
High blood pressure (BP) is a major risk factor for coronary artery disease (CAD), with 30-70% of CAD patients having elevated BP. The conventional method of measuring BP in the arm (brachial BP) may miss some cases, as individuals can have normal brachial pressure but elevated central systolic pressure, which is a more critical predictor of cardiovascular events. Lowering BP is a key objective in cardiac rehabilitation programs.

Examining BP responses after a single bout of exercise could help predict how effectively exercise lowers BP over time. There is a well-established reduction in BP, known as post-exercise hypotension (PEH), which occurs after exercise. This drop is typically around 8 to 9 mmHg and is observed in individuals with and without hypertension. However, it may not occur in people with CAD. The reason for this difference is unclear but may relate to individual variability in exercise responses.

No research has closely examined individual responses to PEH in people with CAD, and it remains unclear whether exercise affects central and brachial BP differently, as some medications do. Additionally, exercise intensity may influence the magnitude of the BP reduction post-exercise. Higher-intensity exercise tends to cause a more significant BP drop, both in hypertensive and non-hypertensive individuals, typically within 20 to 60 minutes post-exercise.

Therefore, the present study aimed to determine the acute effects of combined exercise at different intensities on central and brachial blood pressure in individuals with and without coronary artery disease.

The key research questions were:

1. Is the BP response of central and brachial arteries to acute combined exercise similar? How does coronary artery disease influence these BP responses? Is there individual variability among people with CAD?
2. Does high-intensity exercise, compared to moderate-intensity exercise, produce more pronounced changes in BP in the post-acute exercise period?

All participants were asked to:

Complete two combined exercise sessions - one moderate- and one high-intensity bout. The order of the sessions was randomly assigned, similar to flipping a coin.

BP was measured before and after each acute exercise bout in the laboratory. The researchers compared central and brachial BP responses between exercise intensities (high vs. moderate) and populations (individuals with and without CAD).

DETAILED DESCRIPTION:
This study was designed as a randomized cross-over, repeated measures experiment. All participants underwent two combined exercise sessions of varying intensities, specifically high (HIGH) and moderate (MOD), in a randomized sequence (http://www.randomizer.org/). Before the exercise sessions, all participants underwent both cardiopulmonary exercise testing and 1RM testing, followed by a DEXA scan during a subsequent visit to the laboratory. Each participant completed all experimental sessions consistently at the same time of the day, specifically in the mornings, with at least 48h between sessions to reduce diurnal variation. Post-exercise measurements were conducted at 5, 15 and 30 min after exercise. Participants reported to the laboratory in a fasted state (≥ 4h), and refrained from vigorous exercise, vitamin supplements, and foods/beverages containing caffeine and alcohol for at least 12 h preceding each experimental session.

ELIGIBILITY:
Inclusion criteria for the coronary artery disease group:

* Middle-aged and older adults with stable coronary artery disease (over 55 years old)

Inclusion criteria for the control group:

* Aged-matched healthy adults free of cardiovascular, respiratory, or metabolic disease and with no more than 2 traditional risk factors.
* Physically active defined as engaging in exercise at least 3 times per week over the past 6 months

Exclusion criteria for both groups:

* Cognitive impairment
* Pulmonary disease
* Uncontrolled atrial or ventricular dysrhythmia
* Disability or mental illness
* Extra-cardiac disease

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Central blood pressure | Baseline, before acute combined exercise/applanation tonometry; 5, 15 and 30 minutes after acute combined exercise
  Central systolic blood pressure (cSBP) was measured using non-invasive carotid tonometry (Complior, ALAM Medical) with participants in a supine position. Carotid waveforms were calibrated from brachial diastolic BP (bDBP) and mean arterial pressure (2/3 bDBP + 1/3 bSBP), assumed constant throughout the vascular system. A single operator performed 2 repeated measurements on the right side, each with 10 waveforms of higher than 90% quality, and the average was used. The pressure from wave reflection on SBP was derived as the difference between bSBP and cSBP.
Brachial blood pressure | Baseline, before acute combined exercise/applanation tonometry; 5, 15 and 30 minutes after acute combined exercise
  Brachial Blood pressure was measured in the supine position using an Omron sphygmomanometer after a 10-min rest. Hypertension was defined per ESH guidelines (bSBP ≥140 mmHg and/or bDBP ≥90 mmHg).

SECONDARY OUTCOMES:
Carotid femoral pulse wave velocity (cfPWV) | Baseline, before acute combined exercise/applanation tonometry; 5, 15 and 30 minutes after acute combined exercise
  Central arterial stiffness was measured via carotid-femoral pulse wave velocity (cf PWV), wherein both carotid and femoral waveforms were collected simultaneously using piezoelectric pressure mechanotransducers (Complior, ALAM Medical, Paris, France). Pulse transit times (PTT) were automatically calculated using the intersect tangent algorithm of the foot-to-foot method, enabling the calculation of cfPWV as the ratio of distance to PTT. Travel time distances were defined as the taped measured distance over body surfaces between the two recording sites of interest, with the cf distance corrected by a factor of 0.8.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Motricidade Humana - University of Lisbon, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Data obtained in this study may be provided to qualified researchers with an academic interest in vascular responses to exercise in people with coronary artery disease. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.

REFERENCES:
- [Background] Iellamo F, Perrone MA, Caminiti G, Volterrani M, Legramante JM. Post-exercise Hypotension in Patients With Coronary Artery Disease. Front Physiol. 2021 Dec 22;12:788591. doi: 10.3389/fphys.2021.788591. eCollection 2021. PMID 35002770
- [Background] Kiviniemi AM, Hautala AJ, Karjalainen JJ, Piira OP, Lepojarvi S, Ukkola O, Huikuri HV, Tulppo MP. Acute post-exercise change in blood pressure and exercise training response in patients with coronary artery disease. Front Physiol. 2015 Jan 12;5:526. doi: 10.3389/fphys.2014.00526. eCollection 2014. PMID 25628572
- [Background] Fagard R, Vanhees L. Twenty-four hour blood pressure after exercise in patients with coronary artery disease. J Hum Hypertens. 2000 Apr;14(4):231-4. doi: 10.1038/sj.jhh.1000976. PMID 10805047
- [Derived] Gaspar MP, Maroco JL, Cruz L, Laranjo S, Santa-Clara H, Fernhall B, Melo X. Repeatability of heart-rate variability and baroreflex sensitivity as metrics of cardiac autonomic function during exercise in young females and males. Eur J Appl Physiol. 2025 Oct 25. doi: 10.1007/s00421-025-06011-w. Online ahead of print. PMID 41137920
- [Derived] Maroco JL, Angarten V, Pinto R, Santos V, Fernhall B, Santa-Clara H, Melo X. Post-exercise differential response of central and brachial blood pressure in patients with coronary artery disease: A randomized crossover trial. PLoS One. 2025 Feb 21;20(2):e0317212. doi: 10.1371/journal.pone.0317212. eCollection 2025. PMID 39982938